CLINICAL TRIAL: NCT07383090
Title: The Effect of Mindfulness-Based Education Given to Female University Students on Sexual/Reproductive Health Stigma and Self-Esteem: a Randomized Controlled Study
Brief Title: Mindfulness-Based Education on Sexual/Reproductive Health Stigma and Self-Esteem in Female University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EDA OZYON ETLI (Other)
Responsible Party: Sponsor-Investigator, EDA OZYON ETLI, Lecturer, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21764
Record Dates: First submitted 2026-01-05; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Mindfulness; Sexual Health; Social Stigma; Self Esteem
Keywords: Mindfulness; Sexual/reproductive health; Stigma; Self-esteem; Nursing
MeSH Terms: conditions — Social Stigma; Coitus | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding was applied for the statistician and in the reporting process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Education Group (Experimental): Participants in this group receive a mindfulness-based education program designed to increase awareness related to sexual and reproductive health, reduce stigma, and improve self-esteem. The program is delivered through structured educational sessions conducted over a defined period.
  Interventions: Behavioral: Mindfulness-Based Education Program
- Control Group (No Intervention): Participants in the control group do not receive any intervention and continue with their usual routine during the study period.

INTERVENTIONS:
Behavioral: Mindfulness-Based Education Program — The intervention consists of a 4-week structured mindfulness-based education program. Participants in the experimental group attend one 60-minute session per week. The program covers mindfulness meditation, body scan techniques, and cognitive exercises focused on reducing sexual/reproductive health stigma and enhancing self-esteem
  Other Names: Mindfulness-Based Stress Reduction
  Arms: Mindfulness-Based Education Group

SUMMARY:
This study was conducted to determine the effect of a mindfulness-based education program on mindfulness level, reproductive and sexual health stigma, and self-esteem among young women.

DETAILED DESCRIPTION:
The research was designed as a quasi-experimental pretest-posttest control group study. The experimental group received a 4-week "Mindfulness-Based Education Program" with one session per week. Data were collected using the Personal Information Form, the Mindfulness Scale (MS), the Young Women's Reproductive and Sexual Health Stigma Scale (YWRSHSS), and the Rosenberg Self-Esteem Scale (RSES). Follow-up measurements were conducted one and three months after the training.

ELIGIBILITY:
Inclusion Criteria:

* Female students aged 18 years and older
* Enrolled in a vocational school of health services
* Volunteering to participate in the study
* Fluent in speaking and understanding Turkish

Exclusion Criteria:

* Female students pursuing a second university degree
* Students currently receiving mindfulness training or sexual health education outside of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants are eligible for the study as it focuses on young women's reproductive health stigma
Enrollment: 48 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Change in Mindfulness Attention Awareness Scale (MAAS) Score | Baseline, Post-intervention (4th week), 1st-month follow-up, and 3rd-month follow-up
  Total score from the Mindfulness Attention Awareness Scale. It consists of 15 items. Higher scores indicate higher levels of dispositional mindfulness.
Change in Young Women's Reproductive and Sexual Health Stigma Scale (YWRSHSS) Score | Baseline, Post-intervention (4th week), 1st-month follow-up, and 3rd-month follow-up
  Total score from the Young Women's Reproductive and Sexual Health Stigma Scale. It consists of 20 items. Scores range from 0 to 20, where higher scores indicate higher levels of perceived stigma
Change in Rosenberg Self-Esteem Scale (RSES) Score | Baseline, Post-intervention (4th week), 1st-month follow-up, and 3rd-month follow-up
  Total score from the Rosenberg Self-Esteem Scale (Short Form). It consists of 20 items assessing self-worth. Higher scores represent more positive self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Emel E EGE, Prof. Dr., Principal Investigator — Necmettin Erbakan University
Locations (1):
- Istanbul Beykent University., Istanbul, Beylikduzu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this study may be shared with researchers upon reasonable request via email to the corresponding author.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after the study results are published and for a period of up to 5 years.
Access Criteria: Researchers must provide a clear research objective and sign a data access agreement.

REFERENCES:
- [Background] Lee SH, Cho SJ. Cognitive Behavioral Therapy and Mindfulness-Based Cognitive Therapy for Depressive Disorders. Adv Exp Med Biol. 2021;1305:295-310. doi: 10.1007/978-981-33-6044-0_16. PMID 33834406
- See also: PubMed — https://pubmed.ncbi.nlm.nih.gov/?term=mindfulness